CLINICAL TRIAL: NCT01501188
Title: Study on the Effect of Kinesio Taping on Bioelectrical Activity of Gastrocnemius Muscles and Range of Ankle Motion in Post-menopausal Women With Chronic Venous Insufficiency
Brief Title: Efficacy Study of Kinesio Taping to Treat Muscular and Joint Problems in Chronic Venous Insufficiency
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Encarnación Aguilar Ferrandiz, Research and teaching staff of the University of Granada, Universidad de Granada
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: UGR-409
Record Dates: First submitted 2011-12-21; First posted 2011-12-29 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Venous Insufficiency
Keywords: Chronic Venous Insufficiency; Kinesio Taping; Electromyography; Range of ankle motion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Kinesio taping (Experimental): Specific type of muscle and joint taping
  Interventions: Other: Kinesio Taping
- Kinesio taping placebo (Placebo Comparator): Kinesio taping placebo
  Interventions: Other: Placebo kinesio taping

INTERVENTIONS:
Other: Kinesio Taping — The participants were randomly assigned to an experimental group, to received Kinesio Taping application for gastrocnemius muscle enhancement and functional correction of the ankle.The treatment was performed three times a week during a 4-week period.
  Other Names: Neuromuscular tape
  Arms: Kinesio taping
Other: Placebo kinesio taping — Placebo-control group received treatment with a sham Kinesio Taping protocol to enhance gastrocnemius muscle function and dorsal ankle flexion.The strips used in this group did not follow the principles of tension and anatomic distribution of Kinesio technique.The treatment was performed three times a week during a 4-week period
  Other Names: Neuromuscular taping placebo
  Arms: Kinesio taping placebo

SUMMARY:
The purpose of this study is to analyze the effects of Kinesio Taping on gastrocnemius muscle activation during gait and on Range of ankle motion in postmenopausal females with Chronic Venous Insufficiency in initial stages in comparison to a placebo control group.

DETAILED DESCRIPTION:
Chronic Venous Insufficiency (CVI) is a very common disease. Patients with this pathology present peripheral muscle pump impairment and restricted range of ankle motion. Few data are available on the use in chronic venous insufficiency patients of Kinesio Taping, a physical therapist's elastic dressing that permits action on muscle activity and joint range.

ELIGIBILITY:
Inclusion Criteria:

* Age between 50 and 75 years.
* Mild-moderate Chronic Venous Insufficiency (grades C1, C2, and C3 on clinical-etiologic-anatomic-pathophysiologic (CEAP) scale)

Exclusion Criteria:

* Chronic Venous Insufficiency (> grade C3)
* Arterial disorders
* Cardiorespiratory disease
* Contraindications for Kinesio Taping technique including thrombosis, wounds, severe trauma, generalized edema secondary to cardiac or renal problems, carcinomas, intolerability of/allergy to surgical tape and pregnancy.

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2008-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Change on surface electromyography in gastrocnemius muscles | At baseline and 4 weeks.
  Muscle activity data during gait is sampled at 1600 Hz by surface electromyography, applying electrodes at medial gastrocnemius and lateral gastrocnemius level in both legs. We follow Surface ElectroMyoGraphy for the Non-Invasive Assessment of Muscles (SENIAM) guidelines for electrode placement and signal processing methods. The patient is instructed on the gait speed. After setting the speed-metronome, the electromyography image and activity is recorded for a total of seven seconds and expressed in microvolts units
Change on range of ankle motion | Baseline and 4 weeks
  This variable is measured by using a digital goniometer(SG 110, Penny and Giles Biometrics Ltd;UK) during maximum dorsal and plantar flexion.A sensor is placed at 10 cm from the internal malleolus and another on the inner side of the foot, parallel to the axial axis and perpendicular to the tibial axis.The machine records the degrees of plantar and dorsal flexion from the neutral position of the ankle.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Moreno, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- University of Granada, Granada, Granada, Spain